CLINICAL TRIAL: NCT06582342
Title: Is 3-D Imaging Technology Superior to Computed Tomography in Assessing Response to Neoadjuvant Treatment in Patients With Borderline or Locally Advanced Pancreatic Adenocarcinoma?
Brief Title: Is the 3D-PANC MSP Model Superior to CT for Assessing Response to Neoadjuvant Treatment in PCA Patients?
Status: Recruiting | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: 3D-PANC
Record Dates: First submitted 2024-08-27; First posted 2024-09-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Adenocarcinoma of the Pancreas
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case-crossover group: All patients included in the study will undergo preoperative CT (conventional protocol) and 3D-MSP reconstruction. These results will be compared with the results of the surgery and the anatomopathological study. Each patient will be evaluated by both techniques of the study, thus serving as his or her own control.
  Interventions: Procedure: Three dimensional imaging technology (3D-PANC MSP model); Procedure: Computerized tomography group (conventional CT)

INTERVENTIONS:
Procedure: Three dimensional imaging technology (3D-PANC MSP model) — The processing of the CT images obtained in each center for the creation of the 3D model will be performed centrally by the team of radiologists and computer scientists of the company Cella Medical Solutions. This team will be blinded to the reports of the CT scans.For each patient 4 NCCN check-lists will be filled in without knowing the result of the surgery or the AP study: 2 based on the conventional CT and two based on the 3D-MSP study.
Procedure: Computerized tomography group (conventional CT) — A multiphase CT (venous phase and pancreatographic phase) with 1mm thick slices and series of images in coronal, axial and sagittal reconstructions will be performed. This CT model will be performed at disease diagnosis and after completion of neoadjuvant chemotherapy treatment. Both CT scans will be independently reported by a radiologist from the hospital of origin. The preoperative CT scan will also be evaluated a posteriori by a radiologist from the sponsoring center with expertise in PAC. Both reports (the one from the radiologist of the center and the one from the radiologist of the sponsoring center) will be used to fill out the imaging study variables sheet based on the latest version of the NCCN 2022 guidelines. The radiologists will not know the outcome of the surgery or the anatomic pathology study at the time of the completion of the report.

SUMMARY:
Prospective multicenter study in which all patients with borderline or locally advanced pancreatic adenocarcioma undergoing neoadjuvant chemotherapy and surgical exploration with curative intent will be included for one year. Preoperative images by traditional CT and 3D-MSP technology will be evaluated, comparing the accuracy variables (sensitivity, specificity, predictive values, area under the curve, concordance index) of both techniques with the gold standard (results of surgery and histopathological analysis).

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy followed by surgery represents the treatment of choice for patients with borderline and locally advanced pancreatic adenocarcinoma (PAC). Despite being the diagnostic technique of choice for PAC staging, computed tomography (CT) has a very low accuracy in detecting those patients who may benefit from surgical resection after neoadjuvant chemotherapy. Consequently, the study of computerized image processing technologies is gaining importance. However, there are no prospective validation studies of these technologies to determine their usefulness in the preoperative evaluation of PCA patients undergoing neoadjuvant therapy.

A prospective multicenter study in which all patients with borderline or locally advanced PAC undergoing neoadjuvant chemotherapy and surgical exploration with curative intent will be included for one year. Preoperative images by traditional CT and 3D-MSP technology will be evaluated, comparing the accuracy variables (sensitivity, specificity, predictive values, area under the curve, concordance index) of both techniques with the gold standard (results of surgery and histopathological analysis).

A prospective, multicenter study with control group will be performed. Since this is the evaluation of a diagnostic test, it will not be necessary to randomize the patients included, since each patient will be evaluated by means of both techniques under study, thus serving as his or her own control.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a diagnosis of borderline or locally advanced PAC of the head of the pancreas, as defined by the National Comprehensive Cancer Network (NCCN), who have received neoadjuvant treatment and who undergo surgical exploration with resective intent.

Exclusion Criteria:

* Patients younger than 18 years of age.
* Patients under 18 years of age.
* Disease progression during neoadjuvant treatment.
* No preoperative CT scan.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of borderline or locally advanced PAC of the head of the pancreas who have received neoadjuvant treatment in Spanish hospitals with extensive experience in the treatment of patients with adenocarcinoma of the pancreas and who are part of the pancreatic surgery research group.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To compare the accuracy of the 3D-MSP model versus conventional CT for preoperative diagnosis of vascular involvement (venous and/or arterial) after neoadjuvant chemotherapy in patients with borderline or locally advanced PCA. | Through study completion, an average of 2 months
  Vascular (arterial and/or venous) involvement by the tumor. The sensitivity, specificity, predictive values and area under the ROC curve of the preoperative evaluation by conventional CT and 3D-MSP model will be compared with the result of the surgery and the pathological anatomy of the tumor (gold standard).

SECONDARY OUTCOMES:
To analyze the accuracy of 3D-MSP technology in evidencing response to neoadjuvant chemotherapy. | Through study completion, an average of 2 months
  The sensitivity, specificity, predictive values and area under the ROC curve of the preoperative evaluation by conventional CT and 3D-MSP model will be compared with the result of the surgery and the pathological anatomy of the tumor (gold standard).
To determine whether quantitative texture analysis (radiomics) has a higher sensitivity and specificity than CT for diagnosing vascular involvement (venous and/or arterial) in the study group. | Through study completion, an average of 2 months
  A posteriori, a texture analysis will be performed on both tumor tissue and adjacent tissue by Cella's radiomics team. Approximately 1500 features related to intensity (histogram), shape (volume), transform-based and radial descriptors will be extracted.
Validate the usefulness of 3D-MSP technology for application in teaching, patient communication and surgical planning. | Through study completion, an average of 2 months
  A multi-question, multi-response survey will be used to subjectively determine the usefulness of the 3D model. The surveys will be answered by expert pancreatic surgeons and residents who did not participate and who are unfamiliar with the outcome of the surgery and the pathological anatomy. We will evaluate 3 areas of of interest: anatomy, surgical planning, and teaching. The ability of the 3D model for patient-physician communication will also be explored. Patients visualize the traditional CT images and the 3D model after surgery by

CONTACTS AND LOCATIONS:
Locations (17):
- Spain (17):
  - Hospital General de Alicante, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital del Mar (Barcelona), Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital German Trias y Puyol, Barcelona
  - Hospital Nuestra señora de la Candelaria, Candelaria
  - Hospital General de Castellón, Castellon
  - Hospital Carlos Haya, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Son Espases Palma de Mallorca, Palma de Mallorca
  - Hospital Virgen del Rocío, Seville
  - Hospital Juan XXIII Tarragona, Tarragona
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Dr Peset, Valencia
  - Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No